CLINICAL TRIAL: NCT04088981
Title: Physicians Committee for Responsible Medicine, A Randomized, Crossover Trial of the Effect of a Dietary Intervention on Intracellular Lipid, Insulin Sensitivity, and Glycemic Control in Type 2 Diabetes
Brief Title: Effect of a Dietary Intervention on Intracellular Lipid Levels, Insulin Sensitivity, and Glycemic Control in Type 2 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not initiated due to COVID-19 restrictions during the original study start date. After the restrictions were lifted, the study was redesigned and entered as a different study.
Sponsor: Physicians Committee for Responsible Medicine (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00037991
Record Dates: First submitted 2019-09-06; First posted 2019-09-13 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: insulin sensitivity; glycemic control; intramyocellular; nutrition; hepatocellular
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: randomized, cross-over
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-fat, vegan diet (Active Comparator): For a 22-week period, participants will be asked to follow a low-fat vegan diet which consists of whole grains, vegetables, legumes, and fruits, with no restriction on energy intake. Animal products and added oils will be excluded. In choosing grain products and starchy vegetables (e.g., bread, potatoes), participants will be encouraged to select those retaining their natural fiber and having a glycemic index <70, using tables standardized to a value of 100 for glucose.
  Interventions: Behavioral: Dietary intervention
- Portion-controlled diet (Active Comparator): For a 22-week period, participants will be asked to follow a portion-controlled diet which will include individualized diet plans that reduce daily energy intake by 500 kcal for overweight participants, and keep carbohydrate intake reasonably stable over time. It will derive 50% of total energy from carbohydrates, 20% from protein, and less than 30% from fat (≤7% saturated fat), with less than 200 mg/day of cholesterol/day.
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Behavioral: Dietary intervention — Low-fat, plant-based diet and a portion-controlled diet

SUMMARY:
The purpose of this study is to compare the effects of a low-fat, plant-based dietary intervention and a portion-controlled dietary intervention (compliant with current American Diabetes Association (ADA) guidelines) on changes in intramyocellular and hepatocellular lipid content in adults with type 2 diabetes. Changes in insulin sensitivity and glycemic control will also be assessed in this study. The study duration is 44 weeks.

DETAILED DESCRIPTION:
Type 2 diabetes is a disease characterized by discordance between the amount of insulin produced by pancreatic β-cells and the amount of insulin required to overcome insulin resistance in the liver and peripheral tissues. The development of insulin resistance has been strongly associated with the prolonged accumulation of lipids (fats) in the liver cells ("hepatocellular lipid") and muscle cells ("intramyocellular lipid"). Conventional pharmacologic therapeutics for type 2 diabetes, like metformin, are designed to reduce the accumulation of hepatocellular and intramyocellular lipids and, thereby, augment insulin sensitivity. Research has shown that a low-fat, plant-based diet, in which the consumption of lipids is limited, is a similarly effective therapeutic intervention for the reduction of hepatocellular and intramyocellular lipid content and the improvement of insulin sensitivity in type 2 diabetes.

The purpose of this study is to compare the effects of low-fat, plant-based dietary intervention and a portion-controlled dietary intervention (compliant with current American Diabetes Association (ADA) guidelines) on hepatocellular and intramyocellular lipid content in adults with type 2 diabetes. Using a cross-over design, participants with type 2 diabetes will be randomly assigned to start with a plant-based or a portion-controlled diet for 22 weeks. The two groups will then switch to the opposite diet regimen for an additional 22 weeks. Before and after each intervention period, the investigators will measure intramuscular and liver fat content. The investigators will also assess the relationship between these variables, insulin sensitivity, and glycemic control.

The investigators hypothesize that both dietary interventions will result in reductions in intramuscular and liver fat content, and that these changes will be associated with improvements in insulin sensitivity and glycemic control in individuals with type 2 diabetes. The investigators further hypothesize that the low-fat, plant-based dietary intervention will elicit greater changes in intracellular lipid concentration, compared with the portion-controlled dietary intervention.

ELIGIBILITY:
Inclusion criteria are as follows:

1. Men and women with type 2 diabetes treated by diet and/or oral hypoglycemic agents other that sulfonylureas
2. Age ≥18 years
3. Body mass index 26-40 kg/m2
4. Medications (antidiabetic, antihypertensive, and lipid-lowering) have been stable for the past 3 months
5. HbA1c between 6-10.5% (42-88 mmol/mol)

Exclusion criteria are as follows:

1. Diabetes mellitus, type 1 and/or treatment with insulin or sulfonylureas
2. Metal implants, such as a cardiac pacemaker or an aneurysm clip
3. History of any endocrine condition that would affect body weight, such as thyroid disease, pituitary abnormality, or Cushing's syndrome
4. Smoking during the past six months
5. Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
6. Use of recreational drugs in the past 6 months
7. Use within the preceding six months of medications that affect appetite or body weight, such as estrogens or other hormones, thyroid medications, systemic steroids, antidepressants (tricyclics, MAOIs, SSRIs), antipsychotics, lithium, anticonvulsants, appetite suppressants or other weight-loss drugs, herbs for weight loss or mood, St. John's wort, ephedra, beta blockers
8. Pregnancy or intention to become pregnant during the study period
9. Unstable medical or psychiatric illness
10. Evidence of an eating disorder
11. Likely to be disruptive in group sessions
12. Already following a low-fat, vegan diet
13. Lack of English fluency
14. Inability to maintain current medication regimen
15. Inability or unwillingness to participate in all components of the study
16. Intention to follow another weight-loss method during the trial

Participants will also review and complete the Yale MRI Safety Questionnaire to determine eligibility for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Intramyocellular lipid content | 1.) Change from week 0 to week 22; 2.) Change from week 22 to week 44
  Proton magnetic resonance (MR) spectroscopy at 4T (Bruker) will be implemented to quantify intramyocellular lipid concentrations.
Hepatocellular lipid content | 1.) Change from week 0 to week 22; 2.) Change from week 22 to week 44
  Proton magnetic resonance (MR) spectroscopy at 4T (Bruker) will be implemented to quantify intramyocellular lipid concentrations.
Insulin sensitivity | Change from baseline to 22 weeks and change from 22 weeks to 44 weeks
  Insulin resistance will be assessed by the Homeostatic Model Assessment (HOMA) PREDIM indexes
Concentration of glucose | 1.) Change from week 0 to week 22; 2.) Change from week 22 to week 44
  Concentration of glucose will be assessed during a standard meal test (Boost Plus, Nestle, Vevey, Switzerland; 720 kcal, 34% of energy from fat, 16% protein, 50% carbohydrate). Plasma concentrations of glucose will be measured at 0, 30, 60, 120, and 180 min.
Concentration of C-peptide | 1.) Change from week 0 to week 22; 2.) Change from week 22 to week 44
  Concentration of C-peptide be assessed during a standard meal test (Boost Plus, Nestle, Vevey, Switzerland; 720 kcal, 34% of energy from fat, 16% protein, 50% carbohydrate). Concentration of C-peptide will be measured at 0, 30, 60, 120, and 180 min.
Rate of glycemic control | 1.) Change from week 0 to week 22; 2.) Change from week 22 to week 44
  Rate of glycemic control will be assessed through HbA1C.

SECONDARY OUTCOMES:
Resting energy expenditure | Change from baseline to 22 weeks and change from 22 weeks to 44 weeks
  Resting energy expenditure REE (pulse, respiratory rate and body temperature) will be measured for 20 minutes through indirect calorimetry utilizing a ventilated hood system in fasting participants.
Postprandial metabolism | Change from Baseline to 22 weeks and change from 22 weeks to 44 weeks
  Postprandial metabolism will be measured by indirect calorimetry. Participants will be asked to report to the laboratory within 60 minutes of waking and after a 12-hour fast. Following 30 minutes of quiet rest in a dimly lit room, pulse, respiratory rate, and body temperature will be measured. Resting energy expenditure will be measured for 20 minutes through indirect calorimetry utilizing a ventilated hood system. Postprandial metabolism will be measured four times, 20 minutes each time, over the course of 3 hours after the standard breakfast.
Body Composition | Change from baseline to 22 weeks and change from 22 weeks to 44 weeks
  Body composition will be measured by dual energy x-ray absorptiometry (Lunar iDXA, GE Healthcare; Madison WI), assessing visceral adipose tissue volume and mass.
Gut microbiome composition | Change from baseline to 22 weeks and change from 22 weeks to 44 weeks
  Quantitative determination of microorganisms and global analysis of microbial diversity from stool sample. The mean of the change between time points in bacteria counts.
Concentration of plasma lipids | Change from baseline to 22 weeks and change from 22 weeks to 44 weeks
  Change in plasma cholesterol & triglycerides.
Body weight | Change from baseline to 22 weeks and change from 22 weeks to 44 weeks
  Change in body weight measured on a calibrated scale.

OTHER OUTCOMES:
Advanced Glycation Endproducts (AGEs) | 1.) Change from week 0 to week 22; 2.) Change from week 22 to week 44
  Advanced Glycation Endproducts (AGEs) will be measured using the AGE Reader mu by Diagnoptics.
Endothelial function | 1.) Change from week 0 to week 22; 2.) Change from week 22 to week 44
  Endothelial function will be measured through use of the itamar EndoPAT, which quantifies the endothelium-mediated changes in vascular tone elicited by a 5-minute occlusion of the brachial artery.

CONTACTS AND LOCATIONS:
Overall Officials: Hana Kahleova, MD, PhD, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Upon request individual participant data will be available to other researchers.

REFERENCES:
- [Background] Ferrannini E, Gastaldelli A, Miyazaki Y, Matsuda M, Pettiti M, Natali A, Mari A, DeFronzo RA. Predominant role of reduced beta-cell sensitivity to glucose over insulin resistance in impaired glucose tolerance. Diabetologia. 2003 Sep;46(9):1211-9. doi: 10.1007/s00125-003-1169-6. Epub 2003 Jul 23. PMID 12879253
- [Background] Krssak M, Falk Petersen K, Dresner A, DiPietro L, Vogel SM, Rothman DL, Roden M, Shulman GI. Intramyocellular lipid concentrations are correlated with insulin sensitivity in humans: a 1H NMR spectroscopy study. Diabetologia. 1999 Jan;42(1):113-6. doi: 10.1007/s001250051123. PMID 10027589
- [Background] Perseghin G, Scifo P, De Cobelli F, Pagliato E, Battezzati A, Arcelloni C, Vanzulli A, Testolin G, Pozza G, Del Maschio A, Luzi L. Intramyocellular triglyceride content is a determinant of in vivo insulin resistance in humans: a 1H-13C nuclear magnetic resonance spectroscopy assessment in offspring of type 2 diabetic parents. Diabetes. 1999 Aug;48(8):1600-6. doi: 10.2337/diabetes.48.8.1600. PMID 10426379
- [Background] Shulman GI. Ectopic fat in insulin resistance, dyslipidemia, and cardiometabolic disease. N Engl J Med. 2014 Sep 18;371(12):1131-41. doi: 10.1056/NEJMra1011035. No abstract available. PMID 25229917
- [Background] Goodpaster BH, Theriault R, Watkins SC, Kelley DE. Intramuscular lipid content is increased in obesity and decreased by weight loss. Metabolism. 2000 Apr;49(4):467-72. doi: 10.1016/s0026-0495(00)80010-4. PMID 10778870
- [Background] Sinha R, Dufour S, Petersen KF, LeBon V, Enoksson S, Ma YZ, Savoye M, Rothman DL, Shulman GI, Caprio S. Assessment of skeletal muscle triglyceride content by (1)H nuclear magnetic resonance spectroscopy in lean and obese adolescents: relationships to insulin sensitivity, total body fat, and central adiposity. Diabetes. 2002 Apr;51(4):1022-7. doi: 10.2337/diabetes.51.4.1022. PMID 11916921
- [Background] Thamer C, Machann J, Bachmann O, Haap M, Dahl D, Wietek B, Tschritter O, Niess A, Brechtel K, Fritsche A, Claussen C, Jacob S, Schick F, Haring HU, Stumvoll M. Intramyocellular lipids: anthropometric determinants and relationships with maximal aerobic capacity and insulin sensitivity. J Clin Endocrinol Metab. 2003 Apr;88(4):1785-91. doi: 10.1210/jc.2002-021674. PMID 12679474
- [Background] Machado MV, Ferreira DM, Castro RE, Silvestre AR, Evangelista T, Coutinho J, Carepa F, Costa A, Rodrigues CM, Cortez-Pinto H. Liver and muscle in morbid obesity: the interplay of fatty liver and insulin resistance. PLoS One. 2012;7(2):e31738. doi: 10.1371/journal.pone.0031738. Epub 2012 Feb 16. PMID 22359625
- [Background] Larson-Meyer DE, Newcomer BR, Ravussin E, Volaufova J, Bennett B, Chalew S, Cefalu WT, Sothern M. Intrahepatic and intramyocellular lipids are determinants of insulin resistance in prepubertal children. Diabetologia. 2011 Apr;54(4):869-75. doi: 10.1007/s00125-010-2022-3. Epub 2010 Dec 23. PMID 21181394
- [Background] Wang C, Liu F, Yuan Y, Wu J, Wang H, Zhang L, Hu P, Li Z, Li Q, Ye J. Metformin suppresses lipid accumulation in skeletal muscle by promoting fatty acid oxidation. Clin Lab. 2014;60(6):887-96. doi: 10.7754/clin.lab.2013.130531. PMID 25016691
- [Background] Sanchez-Munoz V, Salas-Romero R, Del Villar-Morales A, Martinez-Coria E, Pegueros-Perez A, Franco-Sanchez JG. [Decrease of liver fat content by aerobic exercise or metformin therapy in overweight or obese women]. Rev Invest Clin. 2013 Jul-Aug;65(4):307-17. Spanish. PMID 24304731
- [Background] Bajaj M, Baig R, Suraamornkul S, Hardies LJ, Coletta DK, Cline GW, Monroy A, Koul S, Sriwijitkamol A, Musi N, Shulman GI, DeFronzo RA. Effects of pioglitazone on intramyocellular fat metabolism in patients with type 2 diabetes mellitus. J Clin Endocrinol Metab. 2010 Apr;95(4):1916-23. doi: 10.1210/jc.2009-0911. Epub 2010 Feb 15. PMID 20157197
- [Background] Phielix E, Brehm A, Bernroider E, Krssak M, Anderwald CH, Krebs M, Schmid AI, Nowotny P, Roden M. Effects of pioglitazone versus glimepiride exposure on hepatocellular fat content in type 2 diabetes. Diabetes Obes Metab. 2013 Oct;15(10):915-22. doi: 10.1111/dom.12112. Epub 2013 May 1. PMID 23574533
- [Background] Marchesini G, Petta S, Dalle Grave R. Diet, weight loss, and liver health in nonalcoholic fatty liver disease: Pathophysiology, evidence, and practice. Hepatology. 2016 Jun;63(6):2032-43. doi: 10.1002/hep.28392. Epub 2016 Jan 22. PMID 26663351
- [Background] Greco AV, Mingrone G, Giancaterini A, Manco M, Morroni M, Cinti S, Granzotto M, Vettor R, Camastra S, Ferrannini E. Insulin resistance in morbid obesity: reversal with intramyocellular fat depletion. Diabetes. 2002 Jan;51(1):144-51. doi: 10.2337/diabetes.51.1.144. PMID 11756334
- [Background] Fabris R, Mingrone G, Milan G, Manco M, Granzotto M, Dalla Pozza A, Scarda A, Serra R, Greco AV, Federspil G, Vettor R. Further lowering of muscle lipid oxidative capacity in obese subjects after biliopancreatic diversion. J Clin Endocrinol Metab. 2004 Apr;89(4):1753-9. doi: 10.1210/jc.2003-031343. PMID 15070941
- [Background] Johansson L, Roos M, Kullberg J, Weis J, Ahlstrom H, Sundbom M, Eden Engstrom B, Karlsson FA. Lipid mobilization following Roux-en-Y gastric bypass examined by magnetic resonance imaging and spectroscopy. Obes Surg. 2008 Oct;18(10):1297-304. doi: 10.1007/s11695-008-9484-0. Epub 2008 Apr 8. PMID 18392897
- [Background] Bachmann OP, Dahl DB, Brechtel K, Machann J, Haap M, Maier T, Loviscach M, Stumvoll M, Claussen CD, Schick F, Haring HU, Jacob S. Effects of intravenous and dietary lipid challenge on intramyocellular lipid content and the relation with insulin sensitivity in humans. Diabetes. 2001 Nov;50(11):2579-84. doi: 10.2337/diabetes.50.11.2579. PMID 11679437
- [Background] Sparks LM, Xie H, Koza RA, Mynatt R, Hulver MW, Bray GA, Smith SR. A high-fat diet coordinately downregulates genes required for mitochondrial oxidative phosphorylation in skeletal muscle. Diabetes. 2005 Jul;54(7):1926-33. doi: 10.2337/diabetes.54.7.1926. PMID 15983191
- [Background] Petersen KF, Dufour S, Morino K, Yoo PS, Cline GW, Shulman GI. Reversal of muscle insulin resistance by weight reduction in young, lean, insulin-resistant offspring of parents with type 2 diabetes. Proc Natl Acad Sci U S A. 2012 May 22;109(21):8236-40. doi: 10.1073/pnas.1205675109. Epub 2012 Apr 30. PMID 22547801